CLINICAL TRIAL: NCT02043015
Title: Comprehensive HIV Prevention Package for MSM in Southern Africa: Pilot Study
Brief Title: Comprehensive HIV Prevention Package for MSM in Southern Africa: Pilot Study (Sibanye Health Project)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Patrick S Sullivan, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB00054863; MP3-1R01A1094575 (Other: Other)
Record Dates: First submitted 2014-01-21; First posted 2014-01-23 (Estimated); Results first posted 2018-01-17 (Actual); Last update posted 2018-09-17 (Actual); Status verified 2018-09

CONDITIONS: HIV
Keywords: voluntary counseling and testing (VCT); couples voluntary counseling and testing (CVCT); pre-exposure prophylaxis (PrEP); homosexuality; male; South Africa
MeSH Terms: conditions — Homosexuality | interventions — Pre-Exposure Prophylaxis; HIV Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Comprehensive HIV prevention services (Other): A comprehensive package of HIV prevention services, including condom choices, Condom-compatible lubricant choices, Couples HIV counseling and testing (CVCT), Staff and provider MSM and LGBT sensitization training, HIV Testing and Risk-reduction counseling, Linkage to care, Pre-exposure prophylaxis with FTC/TDF
  Interventions: Behavioral: Condom choices; Behavioral: Condom-compatible lubricant choices; Behavioral: Couples HIV counseling and testing (CVCT); Drug: Pre-exposure prophylaxis with FTC/TDF; Other: Staff and provider MSM and LGBT sensitization training; Behavioral: HIV Testing and Risk-reduction counseling; Behavioral: Linkage to care

INTERVENTIONS:
Behavioral: Condom choices — Men will receive the condom package that includes an assortment of styles, sizes, features and colors at their baseline visit, and will be able to get more condoms for free at any time after that visit by coming to a study clinic during clinic hours, or during a scheduled study visit.
Behavioral: Condom-compatible lubricant choices — Men will receive condom-compatible lubricant that will include different types of lubricant (e.g., silicone-based) and different packaging (individual sachets or flat, discreet packages) at their baseline study visit, and participants will be able to access enhanced condom-compatible lubricant at any time after that visit by coming to a study clinic during clinic hours, or during a scheduled study visit.
Behavioral: Couples HIV counseling and testing (CVCT) — Participants will be invited to schedule couples voluntary HIV counseling and testing (CVCT) appointments with a clinic counselor at any point after they complete their baseline study visit.
Drug: Pre-exposure prophylaxis with FTC/TDF — For men who meet eligibility criteria, PrEP with Emtricitabine/Tenofovir Disoproxil Fumarate (FTC/TDF) will be made available beginning one month into the study. Men who express interest and meet eligibility criteria at their baseline visit can initiate PrEP at 1 month if they test negative for HIV. For men with extenuating circumstances, whose risk profile changes, of those who become more comfortable with the PrEP intervention through enrollment in the study, PrEP will be available to initiate at the 4 month visit. Men who accept PrEP will be required to have clinic visits, in addition to the regularly scheduled study visits, one month after starting PrEP and at least every 3 months afterward to monitor blood creatinine, AST/ALT and phosphorus levels.
  Other Names: PrEP
Other: Staff and provider MSM and LGBT sensitization training — The training for clinicians will focus on specific sexual health issues for MSM, including taking sexual histories in a non-judgmental way, physical examination techniques including anal examinations, and collection of rectal swabs for STI testing. Trainings will include topics about stigma, sexual identity and coming out, anal sex, STIs, and mental health. Training on LGBT sensitization will be provided for medical providers and staff in target clinics.
Behavioral: HIV Testing and Risk-reduction counseling — Risk-reduction counseling will be provided to all men at baseline and additionally at 3, 6, and 12 month visits, with an additional counseling session for men on PrEP at their initiation visit (either month 1 or 4), their 1-month follow-up visit (either month 2 or 5) and at their 9 month visit. Risk reduction counseling will be client-centered counseling, according to CDC's Fundamentals of HIV Prevention Counseling protocol.
Behavioral: Linkage to care — Men will be linked to needed services including HIV care and treatment for positives identified at baseline or during the study, including antiretroviral medications, and mental health services. At the end of their baseline visit, participants will receive service referral handouts for HIV care and treatment, mental health services, and other resources, as appropriate. Men who test positive for STIs will be treated at the clinic site.

SUMMARY:
The purpose of this study is to evaluate the acceptability and uptake of a combination package of biomedical, behavioral and community-level HIV prevention interventions and services for men who have sex with men (MSM) in South Africa.

DETAILED DESCRIPTION:
Study Design:

This pilot study is a longitudinal cohort study of approximately 100 MSM, with a prospective follow-up period of 1 year for each participant. MSM will be recruited through community events, venues where MSM are known to congregate, online, and by participant referral. Following consent, a baseline visit will include a self-administered baseline survey, a clinical exam including an assessment for circumcision and STIs, and testing for HIV and other sexually transmitted infections (STIs), creatinine, AST/ALT and phosphorus levels, and drug screening.

An HIV prevention package will be offered to participants starting at baseline, which will include condom choices, condom-compatible lubricant choices, risk-reduction counseling, linkage to care, and couples voluntary counseling and testing (CVCT). HIV-negative men can be screened for eligibility for pre-exposure prophylaxis (PrEP) with Emtricitabine/Tenofovir Disoproxil Fumarate (FTC/TDF), which will be made available for eligible men beginning at the 1-month or 4-month study visit. Throughout the study, PEP for men with an exposure at high risk for HIV transmission will be made available.

Men who test positive for HIV at baseline or during the study will be referred and actively linked to appropriate care and treatment services and will continue to be a part of the study. Men who test positive for STIs at baseline or during the study will receive treatment at the study clinic. Participants will complete follow-up visits at 3, 6, and 12 months that will include self-administered behavioral surveys and HIV testing, and STI testing at 6 and 12 months.

Men who are eligible and interested in initiating PrEP can return for a PrEP initiation visit, which will include rapid HIV testing, at two time points: 1 month after enrollment and 4 months after enrollment. Men who initiate PrEP will have additional clinic visits for creatinine, AST/ALT, phosphate, protein and glucose level testing and rapid HIV testing the month following PrEP initiation (month 2 for those initiating PrEP at 1 month and month 5 for those initiating PrEP at 4 months) and every 3 months thereafter. If a participant on PrEP tests positive for HIV, they will discontinue PrEP but continue to be followed for their remaining study visits.

Men who test positive for HIV at follow-up visits will have blood drawn for initial cluster of differentiation 4 (CD4) and HIV viral load testing, and will have CD4 testing at 6 and 12 months and HIV viral load testing at 3, 6, and 12 months. Data on service utilization, condom use, lubricant use, HIV and STI testing outside the study site, and other outcomes will be collected via monthly short message service (SMS) text message surveys during the study period.

Study Population:

The study population will be men aged 18 years and older who self-report that they had anal intercourse with men in the past year, are current residents of the study city, are willing to provide contact information, and have a phone.

Study Size:

The sample will consist of approximately 100 MSM in Cape Town, South Africa. All 100 men will be followed for one year, and approximately 20% of the study population can be HIV-infected at baseline. Additional men who are HIV-positive at baseline will be enrolled in the baseline visit but not followed prospectively, and not counted as part of the 100 men in that study site.

Study Intervention:

The prevention package will be offered throughout the study and will include condom choices with an assortment of styles, sizes and features, condom-compatible lubricant choices with discreet packaging, risk reduction counseling, linkage to care, couples voluntary HIV counseling and testing (CVCT), and PrEP for eligible men beginning one month after enrollment. Condom choices, lubricant choices, and CVCT will be available to participants at drop-in visits at any time.

Throughout the study, post-exposure prophylaxis (PEP) for men with an exposure at high risk for HIV transmission will be available as standard of care.

Community-level interventions will occur through training of health care providers to deliver sexual health services to MSM and lesbian, gay, bisexual, and transgender (LGBT) sensitization, LGBT training for study staff and other staff of the clinical sites, and community mobilization efforts to improve health literacy and uptake of prevention services among MSM.

Study Duration:

Recruitment activities will be conducted for 3 months or until 100 MSM have been recruited. After enrollment, MSM will have a follow-up period of 1 year for each participant.

Primary Objectives:

This study has four primary objectives:

1. Determine acceptability of the HIV prevention package.
2. Determine uptake of individual elements of the HIV prevention package.
3. Determine incidence of HIV, STIs and unprotected anal intercourse (UAI).
4. Understand HIV risk and prevention behaviors among MSM.

Participating Sites:

1. Emory University, Atlanta, Georgia
2. Johns Hopkins Bloomberg School of Public Health, Baltimore, Maryland
3. University of California, Los Angeles, Los Angeles, California
4. Desmond Tutu HIV Foundation, Cape Town, South Africa (Enrollment & Clinic site)

ELIGIBILITY:
Inclusion Criteria:

* Male sex at birth
* Anal sex with another man in the past 12 months
* 18 years of age or older
* Resident of the study city
* Able to complete study instruments, with or without assistance, in English, Xhosa or Afrikaans
* Willing to provide contact information
* Has a phone

Exclusion Criteria:

* Not male sex at birth
* No self-reported anal sex with a man in the past 12 months
* Less than 18 years of age
* Not a resident of the study city
* Plans to move from the study city within the year after enrollment
* Not able to complete study instructions, with or without assistance, in English, Xhosa or Afrikaans
* Not willing to provide contact information
* Does not have a phone

Additional Inclusion and Exclusion Criteria for participants on PrEP:

PrEP Inclusion Criteria:

* Identified as high-risk for HIV by the provider by meeting one or more of the criteria below:
* Have multiple partners
* Engage in transactional sex, including sex workers
* Use or abuse drugs
* Drink alcohol heavily
* Had more than 1 episode of a STI in the last year
* Is the HIV-negative partner in a discordant relationship, especially if the HIV-positive partner is not on antiretroviral therapy (ART)
* Is in a non-monogamous concordant relationship with a HIV-negative partner
* Is unable or unwilling to achieve consistent use of male condoms
* No contra-indications to Emtricitabine/Tenofovir Disoproxil Fumarate (FTC/TDF)
* Calculated creatinine clearance of at least 60 mL/min
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 2 x upper limit of normal (ULN)
* Hepatitis B surface antigen (HBsAg) negative
* Motivated to follow PrEP prescribing guidelines
* Willing to adhere to daily oral dosing
* Willing to attend PrEP maintenance visits every 3 months

PrEP Exclusion Criteria:

* HIV positive
* Signs or symptoms suggestive of acute HIV infection
* Have baseline creatinine clearance <60 ml/min
* Are unwilling to follow PrEP prescribing guidelines
* Are unwilling to attend PrEP maintenance visits every 3 months
* Are known to have hypertensives or diabetes
* Are hepatitis B susceptible (test HBsAg and HBsAb negative) and refuse to take a hepatitis B vaccine series
* Any contraindication to taking FTC/TDF
* Proteinuria 2+ or greater at screening
* Glucosuria 2+ or greater at screening
* Use of antiretroviral (ARV) therapy (e.g., for PEP or PrEP) in the 90 days prior to study entry

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick S Sulivan, DVM, PhD, Principal Investigator — Rollins School of Public Health; A.D. McNaghten, PhD, MHSA, Principal Investigator — Rollins School of Public Health; Stefan Baral, MD, MPH, Principal Investigator — Johns Hopkins Bloomberg School of Public Health; Linda-Gail Bekker, MBChB, PhD, Principal Investigator — Desmond Tutu HIV Foundation; Rob Stephenson, MSc, PhD, Principal Investigator — Rollins School of Public Health; Chris Beyrer, MD, MPH, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (3):
- United States (2):
  - Rollins School of Public Health, Atlanta, Georgia
  - Johns Hopkins School of Public Health, Baltimore, Maryland
- Desmond Tutu HIV Foundation, Cape Town, South Africa

REFERENCES:
- [Derived] McNaghten A, Kearns R, Siegler AJ, Phaswana-Mafuya N, Bekker LG, Stephenson R, Baral SD, Brookmeyer R, Yah CS, Lambert AJ, Brown B, Rosenberg E, Blalock Tharp M, de Voux A, Beyrer C, Sullivan PS. Sibanye Methods for Prevention Packages Program Project Protocol: Pilot Study of HIV Prevention Interventions for Men Who Have Sex With Men in South Africa. JMIR Res Protoc. 2014 Oct 16;3(4):e55. doi: 10.2196/resprot.3737. PMID 25325296

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited in Cape Town, South Africa between February 2015 and September 2015. Each participant was followed for one year.
Pre-assignment Details: To obtain the target enrollment of 80 HIV-negative and 20 HIV-positive participants, additional HIV-positive persons consented to participate but were not prospectively followed after the baseline visit. Fifteen participants were study stopped after baseline and not eligible for prospective follow-up to reach the target enrollment numbers.
Groups:
- Recipients of HIV Prevention Services: Study participants receiving a comprehensive package of HIV prevention services including: condom choices, condom-compatible lubricant choices, couples HIV counseling and testing (CVCT), men who have sex with men (MSM) and lesbian, gay, bisexual, and transgender (LGBT) sensitization training for staff and providers, HIV testing, risk-reduction counseling, linkage to care, and pre-exposure prophylaxis with emtricitabine/tenofovir disoproxil fumarate (FTC/TDF).
Period: Overall Study
Arm/Group | Recipients of HIV Prevention Services
Started | 115
Completed | 87
Not Completed | 28
Not completed — Lost to Follow-up | 4
Not completed — Withdrawal by Subject | 4
Not completed — Removed once target enrollment reached | 15
Not completed — Participant moved away from study city | 4
Not completed — Incarceration | 1

BASELINE CHARACTERISTICS:
Population: The Baseline analysis population consists of persons who consented to take part in the study and were eligible to participate.
Groups:
- Recipients of HIV Prevention Services: Study participants receiving a comprehensive package of HIV prevention services including: condom choices, condom-compatible lubricant choices, couples HIV counseling and testing (CVCT), staff and provider MSM and LGBT sensitization training, HIV testing, risk-reduction counseling, linkage to care, and pre-exposure prophylaxis with FTC/TDF.
Arm/Group | Recipients of HIV Prevention Services
Number analyzed (Participants) | 115
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 115
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.3 (7.4)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Eligible participants were male at birth. As part of demographic assessments, all participants were asked to self-identify their gender as Male, Female, Transgender, or Other.
  Participants
    Gender identification: Female | 7
    Gender identification: Male | 99
    Gender identification: Transgender | 5
    Gender identification: Other | 1
    Gender identification: Unknown or not reported | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — As part of demographic assessments, all participants were asked to self-identify their race as Black African, Coloured (a multiracial ethnic group in South Africa), Indian or Asian, White, or Other.
  Participants
    Black African | 89
    Coloured | 21
    White | 4
    Unknown or not reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  South Africa | 115
HIV Status at Baseline Visit [Count of Participants; unit: Participants]
  HIV-Positive at Baseline | 35
  HIV-Negative at Baseline | 80

OUTCOME MEASURES:

1. Primary Outcome: Retention in the Cohort
Description: The ability of the study to retain participants for full study period was assessed. Retention was measured by the number and percentage of enrolled participants attending study visits through the 12-month study period.
Time Frame: 12 months
Population: This analysis includes all participants enrolled for prospective follow-up at baseline. Twenty of the participants tested HIV-positive at baseline, and the remaining 80 tested HIV-negative.
Measure: Count of Participants; unit: Participants
Groups:
- Recipients of HIV Prevention Services: Men receiving a comprehensive package of HIV prevention services including: condom choices, condom-compatible lubricant choices, couples HIV counseling and testing (CVCT), staff and provider MSM and LGBT sensitization training, HIV testing, risk-reduction counseling, linkage to care, and Pre-exposure prophylaxis with FTC/TDF
Arm/Group | Recipients of HIV Prevention Services
Number analyzed (Participants) | 100
Participants
  Participants attending the Month 3 Visit | 88
  Participants attending the Month 6 Visit | 84
  Participants attending the Month 12 Visit | 87

2. Primary Outcome: Use of PrEP
Description: Uptake of PrEP by study participants was measured as the number and percentage of enrolled participants eligible for PrEP at the baseline and 3-month study visits who choose to initiate PrEP at a visit one month later.
Time Frame: 4 months
Population: Of the 80 participants who were HIV-negative at the baseline visit, 60 were PrEP-eligible based on behavioral and clinical criteria. At the Month 3 visit, participants who were not already on PrEP could be assessed for PrEP eligibility again. Participants could be counted as PrEP-eligible at both the Baseline and Month 3 time points.
Measure: Count of Participants; unit: Participants
Arm/Group | Recipients of HIV Prevention Services
Number analyzed (Participants) | 60
Participants
  PrEP Uptake at Month 1 Visit: number analyzed (Participants) | 51
  PrEP Uptake at Month 1 Visit | 39
  PrEP Uptake at Month 4 Visit: number analyzed (Participants) | 11
  PrEP Uptake at Month 4 Visit | 6

3. Primary Outcome: Number of Participants With New HIV Infection
Description: Incident HIV infection is measured as the number of seroconversions during follow-up among those who are HIV-uninfected at baseline.
Time Frame: 12 months
Population: The population includes all participants who were HIV-negative at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Recipients of HIV Prevention Services
Number analyzed (Participants) | 80
Participants | 6

4. Secondary Outcome: Condom Use
Description: Condom use is measured as the number of male anal sex partners that the study participant always used condoms with in the prior three or six months, as self-reported reported in the questionnaire at each study visit.
Time Frame: Months 3, 6, and 12
Population: This analysis includes all participants enrolled for prospective follow-up at baseline.
Measure: Count of Units; unit: Sex partners
Units Other Than Participants: Sex partners
Arm/Group | Recipients of HIV Prevention Services
Number analyzed (Participants) | 100
Number analyzed (Sex partners) | 120
Sex partners
  Month 3 Visit: number analyzed (Participants) | 57
  Month 3 Visit | 84
  Month 6 Visit: number analyzed (Participants) | 55
  Month 6 Visit: number analyzed (Sex partners) | 113
  Month 6 Visit | 82
  Month 12 Visit: number analyzed (Participants) | 52
  Month 12 Visit: number analyzed (Sex partners) | 118
  Month 12 Visit | 84

5. Secondary Outcome: Lubricant Use
Description: Measured as the number and percentage of participants who used condom-compatible lubricant during their most recent anal sex act, among those who also used a condom at their most recent anal sex act.
Time Frame: Months 3, 6, and 12
Population: This analysis includes all participants enrolled for prospective follow-up at baseline who self-reported using a condom during their most recent anal sex reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Recipients of HIV Prevention Services
Number analyzed (Participants) | 53
Participants
  Month 3 Visit: number analyzed (Participants) | 29
  Month 3 Visit | 17
  Month 6 Visit: number analyzed (Participants) | 27
  Month 6 Visit | 14
  Month 12 Visit: number analyzed (Participants) | 21
  Month 12 Visit | 9

6. Secondary Outcome: Voluntary Counseling and Testing (VCT) and Couples Voluntary Counseling and Testing (CVCT) Uptake
Description: VCT and CVCT is measured as the number and percentage of participants who completed VCT in the study period as part of the study visits and the number and percentage of participants who self-reported VCT outside of their study visits. These are compared to the number and percentage of participants who self-reported having VCT in the year prior at baseline. CVCT is measured as the number and percentage of participants who completed a CVCT session as part of the study.
Time Frame: 12 months
Population: Participants who tested HIV-negative at baseline and were enrolled for prospective follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Recipients of HIV Prevention Services
Number analyzed (Participants) | 80
Participants
  VCT during 12 months preceding the study period | 57
  VCT as part of the study | 76
  VCT outside of the study (during study period) | 53
  CVCT during the study period | 1

7. Secondary Outcome: Number of HIV Tests During Study
Description: The number of HIV tests per participant administered during the study period.
Time Frame: 12 months
Population: This analysis includes all participants enrolled for prospective follow-up at baseline.
Measure: Mean (Standard Deviation); unit: HIV tests
Arm/Group | Recipients of HIV Prevention Services
Number analyzed (Participants) | 100
HIV tests | 4.9 (3.0)

8. Secondary Outcome: Serodiscordant Unprotected Anal Intercourse (UAI)
Description: Measured as any self-reported unprotected anal intercourse in the last three or six months with a partner of opposite or unknown HIV status, as self-reported in the questionnaire at each study visit.
Time Frame: Month 3, 6, and 12
Population: The analysis population includes all prospectively followed participants who completed the survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Recipients of HIV Prevention Services
Number analyzed (Participants) | 100
Participants
  Month 3 Visit: number analyzed (Participants) | 85
  Month 3 Visit | 11
  Month 6 Visit: number analyzed (Participants) | 83
  Month 6 Visit | 5
  Month 12 Visit: number analyzed (Participants) | 80
  Month 12 Visit | 4

9. Secondary Outcome: Acceptability of Post-exposure Prophylaxis (PEP)
Description: Measured as the number of men who report an eligible exposure who accept and initiate PEP.
Time Frame: 12 months
Population: Participants who tested HIV-negative at baseline and were followed prospectively.
Measure: Count of Participants; unit: Participants
Arm/Group | Recipients of HIV Prevention Services
Number analyzed (Participants) | 80
Participants | 0

10. Secondary Outcome: Acceptability of Provider Training
Description: Measured as the number of providers who accept the training related to MSM-specific healthcare.
Time Frame: 12 months
Population: The mandatory MSM-specific training had already been completed for health care providers in Cape Town, thus the training specified by the study protocol was no longer necessary.
Groups:
- Health Care Providers: Health care providers in Cape Town who care for MSM populations.
Arm/Group | Health Care Providers
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the entire 12 month study period.
Description: All symptoms reported as possibly or probably related to a study intervention are reported as adverse events. In this study, the interventions include the HIV prevention interventions (condoms, lubricant, CVCT, PrEP) and community interventions. Possible adverse events include social harms such as stigma and discrimination in health care settings, verbal abuse, relationship disruption, and loss of access to services.
Arm/Group | Recipients of HIV Prevention Services
All-Cause Mortality (participants affected / at risk) | 0/100
Serious Adverse Events (participants affected / at risk) | 2/100
Other Adverse Events (participants affected / at risk) | 20/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Recipients of HIV Prevention Services (N=100)
Elevated liver enzymes, secondary to Hepatitis C diagnosis (Hepatobiliary disorders) | 1 (1)
Elevated liver enzymes (Hepatobiliary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Recipients of HIV Prevention Services (N=100)
Fatigue, possibly or probably related to PrEP (General disorders) | 4 (4)
Gastrointestinal symptoms, possibly or probably related to PrEP (Gastrointestinal disorders) | 7 (8)
Thirst, possibly or probably related to PrEP (General disorders) | 2 (2)
Sweating, possibly or probably related to PrEP (General disorders) | 1 (1)
Hypersomnia, possibly or probably related to PrEP (General disorders) | 1 (1)
Hypersensitivity reaction, possibly or probably related to PrEP (Immune system disorders) | 1 (1)
Symptoms of hyperglycemia, possibly or probably related to PrEP (Metabolism and nutrition disorders) | 1 (1)
Hypertension, possibly or probably related to PrEP (Vascular disorders) | 1 (1)
Polydypsia, possibly or probably related to PrEP (General disorders) | 1 (1)
Generalized pruritis, possibly or probably related to PrEP (Skin and subcutaneous tissue disorders) | 1 (1)
Glycosuria, possibly or probably related to PrEP (General disorders) | 1 (1)
Hypersensitivity reaction, possibly or probably related to Hepatitis B vaccination (Immune system disorders) | 1 (1)
Gastrointestinal symptoms, possibly or probably related to sexually transmitted infection treatment (Gastrointestinal disorders) | 1 (1)
Social harm: participant's family member found their PrEP study medication (Social circumstances) | 3 (3)
Dry mouth, possibly or probably related to PrEP (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes